CLINICAL TRIAL: NCT04941950
Title: A Digital Intervention to Prevent the Initiation of Opioid Misuse in Adolescents in School-based Health Centers (Randomized Controlled Trial)
Brief Title: A Digital Intervention to Prevent the Initiation of Opioid Misuse in Adolescents in School-based Health Centers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trustees of Dartmouth College (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2000030553; 1UG3DA050251-01 (NIH)
Record Dates: First submitted 2021-06-23; First posted 2021-06-28 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Opioid Misuse
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PlaySmart (Experimental): Video game intervention.
  Interventions: Behavioral: PlaySmart
- Control Game (Other): Control video game intervention.
  Interventions: Other: Video Game Control

INTERVENTIONS:
Behavioral: PlaySmart — PlaySmart is designed to provide players with behavioral skills and knowledge through repetitive and engaging videogame play to target adolescent perception of risk of harm from initiating opioid misuse.
  Arms: PlaySmart
Other: Video Game Control — Participants in the control group will play another video game with no intended effect similar to PlaySmart.
  Arms: Control Game

SUMMARY:
The primary hypothesis of this study is that at 3 months, there will be a higher proportion of intervention participants vs. control participants who report greater risk of harm from misuse of prescription opioids AND heroin.

DETAILED DESCRIPTION:
This study's specific aims are to:

Conduct a randomized controlled trial with 532 high-risk adolescents in 10 School Based Health Centers (SBHCs), to compare PlaySmart to attention/time control games, with assessments post- gameplay (6 weeks), and at 3, 6, and 12 months following enrollment to determine if PlaySmart: 1) increases proportion of participants who report a perception of great risk of harm from misuse of opioids at 3 months; and 2) decreases intentions to misuse opioids; 3) increases self-efficacy for refusing opioids; 4) prevents initiation of opioid misuse, at all time-points.

ELIGIBILITY:
Inclusion Criteria:

* Participants must:
* 1) preferably be enrolled in their high school's School-Based Health Center;
* 2) report NOT having engaged in any prior opioid misuse;
* 3) be at "high-risk" based on their report at baseline of past 30-day use of cigarettes, e-cigarettes, Juul, alcohol, marijuana (including synthetics), amphetamine, cocaine, benzodiazepines, ecstasy, bath salts, or any other misuse of non-opioid prescription drugs or use of non-opioid illicit drugs OR have a score of ≥1 on the PHQ-2 OR a score of ≥1 on the GAD-2 (both screening tools used by SBHA);
* 4) be willing to sit for 60 minutes/session to play the game;
* 5) be able to provide assent/parental/guardian consent (if under age 18).

Exclusion Criteria:

* Failure to meet any of the inclusion criteria.

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 533 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Perception of Risk | 3 months
  Perceived risk was measured by the question, "How much do you think people risk harming themselves (physically or in other ways), if they..." try or use a drug. For example, "...try marijuana once or twice." The answer categories are "no risk," "slight risk," "moderate risk," "great risk," and "can't say, drug unfamiliar." Parallel questions refer to using the same drug "occasionally" and "regularly." It is an 8 item, 4-point Likert scale. Total score range from 0-24. Higher scores mean greater perception of risk.
Change in Perception of Risk | Baseline, 6 weeks, 3, 6, and 12 months
  Perceived risk was measured by the question, "How much do you think people risk harming themselves (physically or in other ways), if they..." try or use a drug. For example, "...try marijuana once or twice." The answer categories are "no risk," "slight risk," "moderate risk," "great risk," and "can't say, drug unfamiliar." Parallel questions refer to using the same drug "occasionally" and "regularly." It is an 8 item, 4-point Likert scale. Total score range from 0-24. Higher scores mean greater perception of risk. This outcome will be measured at baseline, after 6 weeks of gameplay, and at 3, 6, and 12 months after baseline.

SECONDARY OUTCOMES:
Change in Intentions to Misuse Opioids (p2P Lab Questions) | Baseline, 6 weeks, 3, 6, and 12 months
  The outcomes will be assessed by determining if there was a change in intentions to misuse opioids from baseline after 6 weeks of gameplay, and at 3, 6, and 12 months after baseline. The self-reported data questions were derived from the Monitoring the Future Study. Each item uses a 5-point scale to assess various facets of opioid misuse.
Change in Self Efficacy for Refusing Opioids (p2P Lab Questions) | Baseline, 6 weeks, 3, 6, and 12 months
  The outcomes will be assessed by determining if there was a change in self-efficacy to refuse offers of opioids from baseline after 6 weeks of gameplay and at 3,6, and 12 months after baseline. This will be collected by self-reported data using questions from a study on preventing drug abuse among adolescents. It is a four-item scale for self-efficacy and relates to adolescent's perceived ability to resist pressure to use substances.
Change in Prevention of Initiation of Opioid Misuse (p2P Lab Questions) | Baseline, 6 weeks, 3, 6, and 12 months
  The outcomes will be assessed by determining if a change in substance use behaviors (including prescription and illicit drugs, tobacco, and alcohol) occurred from baseline after 6 weeks of gameplay, and 3, 6, and 12 months after baseline. Self- reported data will be collected using questions from the Monitoring the Future Study.
Change in Knowledge about opioid misuse and its risks and mental health (p2P Lab Questions) | Baseline, 6 weeks, 3, 6, and 12 months
  The outcomes will be assessed by determining a change in knowledge. Data analysis forthcoming.
Change in Attitudes to Misuse Opioids (p2P Lab Questions) | Baseline, 6 weeks, 3, 6, and 12 months
  The outcomes will be assessed by determining a change in attitudes towards misuse opioids. Data analysis forthcoming.
Change in Perceived Norms About Opioid Misuse (p2P Lab Questions) | Baseline, 6 weeks, 3, 6, and 12 months
  The outcomes will be assessed by determining a change in perceived norms towards misuse opioids. Data analysis forthcoming.
Decision-Making Skills (p2P Lab Questions) | Baseline, 6 weeks, 3, 6, and 12 months
  The outcomes will be assessed by determining a change in decision-making skills. Data analysis forthcoming.
Self-Regulation (Across Time-TRAIT DERS) (p2P Lab Questions) | Baseline
  Data analysis forthcoming.
Self-Regulation (In a specific moment-STATE DERS) (p2P Lab Questions) | Baseline, 6 weeks, 3, 6, and 12 months
  The outcomes will be assessed by determining a change in self-regulation. Data analysis forthcoming.
Help-Seeking Behavior (Past) (p2P Lab Questions) | Baseline, 6 weeks, 3, 6, and 12 months
  The outcomes will be assessed by determining a change in help-seeking behaviors. Data analysis forthcoming.
Help Seeking Behavior (General) (p2P Lab Questions) | Baseline, 6 weeks, 3, 6, and 12 months
  The outcomes will be assessed by determining a change in help-seeking behaviors. Data analysis forthcoming.
Self-Stigma of Seeking Help Scale (p2P Lab Questions) | Baseline, 6 weeks, 3, 6, and 12 months
  The outcomes will be assessed by determining a change in self-stigma of seeking help. Data analysis forthcoming.
Beliefs About Psychological Services (p2P Lab Questions) | Baseline, 6 weeks, 3, 6, and 12 months
  The outcomes will be assessed by determining a change in beliefs about psychological services. Data analysis forthcoming.
Gameplay Experience (p2P Lab Questions) | 6 weeks
  Data analysis forthcoming
Gameplay Usability (p2P Lab Questions) | 6 weeks
  Data analysis forthcoming
Gameplay Engagement (p2P Lab Questions) | 6 weeks
  Data analysis forthcoming
Involvement with Legally Manufactured Opioids (Coordinating Center Questions) | Baseline, 6 weeks, 3, 6, and 12 months
  The outcomes will be assessed by a change in involvement with legally manufactured opioids. Data analysis forthcoming
Involvement with Illegally Manufactured Opioids (Coordinating Center Questions) | Baseline, 6 weeks, 3, 6, and 12 months
  The outcomes will be assessed by a change in involvement with illegally manufactured opioids. Data analysis forthcoming
Involvement with Alcohol (Coordinating Center Questions) | Baseline, 6 weeks, 3, 6, and 12 months
  The outcomes will be assessed by a change in involvement with alcohol. Data analysis forthcoming
Involvement with Marijuana (Coordinating Center Questions) | Baseline, 6 weeks, 3, 6, and 12 months
  The outcomes will be assessed by a change in involvement with marijuana. Data analysis forthcoming
Self-Efficacy (Coordinating Center Questions) | Baseline, 6 weeks, 3, 6, and 12 months
  Data analysis forthcoming
Mental Health (Depression - PHQ-8) (Coordinating Center Questions) | Baseline, 6 weeks, 3, 6, and 12 months
  Data analysis forthcoming
Mental Health (Anxiety - GAD-7) (Coordinating Center Questions) | Baseline, 6 weeks, 3, 6, and 12 months
  Data analysis forthcoming
Experience with Pain (Coordinating Center Questions) | Baseline, 6 weeks, 3, 6, and 12 months
  Data analysis forthcoming
Social Exposure to Substance Misuse (Exposure to Drugs and Alcohol) (Coordinating Center Questions) | Baseline, 6 weeks, 3, 6, and 12 months
  Data analysis forthcoming

CONTACTS AND LOCATIONS:
Overall Officials: Lynn E Fiellin, MD, Principal Investigator — Director, play2PREVENT Lab & Professor, BDS at Geisel School of Medicine at Dartmouth College
Locations (15):
- United States (15):
  - Harding High School, Bridgeport, Connecticut
  - Coginchaug High School, Durham, Connecticut
  - CT River Academy, East Hartford, Connecticut
  - Fairfield College Preparatory School, Fairfield, Connecticut
  - Fitch High School, Groton, Connecticut
  - Hamden High School, Hamden, Connecticut
  - Weaver High School, Hartford, Connecticut
  - Maloney High School, Meriden, Connecticut
  - Platt High School, Meriden, Connecticut
  - Hopkins High School, New Haven, Connecticut
  - New London High School, New London, Connecticut
  - Stamford High School, Stamford, Connecticut
  - Westhill High School, Stamford, Connecticut
  - Academy of Information, Technology, and Engineering, Stamford, Connecticut
  - West Haven High School, West Haven, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
The plan will comply with the NIH HEAL Initiative ClinicalTrials.govSM Public Access and Data Sharing Policy, NIH Data Sharing Policy, NIH Policy on Dissemination of NIH-Funded Clinical Trial Information, and NIH Clinical Trial Registration and Results Information Submission rule. All IPD will be in a repository supported by NIDA, the NAHDAP, following NIH requirements for sharing data via creation of public-use data sets. Data will be de-identified/masked to minimize risk of potential re-identification to participants. This may include modification of the original data to reduce risk of re-identification of participants. A structured process will evaluate the risk of re-identification based on guidance documents from the US DHHS, HIPAA, and quantitative evaluation of the data using statistical methods. Potential revisions to the data to prepare them for NAHDAP include omission of variables, collapsing of categories of a variable, or other coarsening of specific participants' values.
Supporting Information: Study Protocol, SAP
Time Frame: HEAL Prevention Cooperative (HPC) data is anticipated to be archived in May 2026.
Access Criteria: The HEAL Coordinating Center will provide HPC data as well as supporting documentation for the HPC Common Measures as well as data that are uniquely collected as part of each HPC Research Project. The NAHDAP repository disseminates data to users based on its Access Policy Framework. Researchers who are not part of the HCP will be able to download HPC datasets and analyze them on their own computers. Access to data requires submission of username, institution, and analytic purpose and aim. There is no formal approval process initially planned by NIDA. Data users are expected to adhere to norms for responsible use.

REFERENCES:
- [Derived] Boomer T, Hoerner L, Larkin K, Maciejewski K, Kyriakides TC, Fiellin LE. A videogame for perceived risk of harm from opioid misuse in adolescents: a randomized controlled trial. Nat Health. 2026;1(1):78-89. doi: 10.1038/s44360-025-00010-z. Epub 2025 Dec 1. PMID 41635738
- [Derived] Pendergrass Boomer TM, Hoerner LA, Fernandes CF, Maslar A, Aiudi S, Kyriakides TC, Fiellin LE. A digital health game to prevent opioid misuse and promote mental health in adolescents in school-based health settings: Protocol for the PlaySmart game randomized controlled trial. PLoS One. 2023 Sep 8;18(9):e0291298. doi: 10.1371/journal.pone.0291298. eCollection 2023. PMID 37683047